CLINICAL TRIAL: NCT00528034
Title: Lymphoscintigraphy and Selective Lymphatic Mapping in Patients With Invasive Vaginal Cancer
Brief Title: Lymphoscintigraphy in Patients With Vaginal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ID02-239
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Vaginal Cancer
Keywords: Vaginal Cancer; Lymphoscintigraphy; Lymphatic Mapping; Sentinel Lymph Node; Isosulfan Blue; Lymph
MeSH Terms: conditions — Vaginal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphoscintigraphy (Experimental)
  Interventions: Procedure: Lymphoscintigraphy

INTERVENTIONS:
Procedure: Lymphoscintigraphy — Procedure where a very small amount (less than one tenth of a teaspoon) of a radioactive material is injected around the edge of the tumor in the vagina, followed immediately by the scan. The scan is done before the patient has surgery or begins radiation therapy.

SUMMARY:
Primary Objectives:

1. Determine the feasibility of using pretreatment lymphoscintigraphy to identify the sentinel lymph node(s) in patients with vaginal cancer dispositioned to receive radiation therapy.
2. Determine the feasibility of using preoperative lymphoscintigraphy and intraoperative lymphatic mapping to identify the sentinel lymph node(s) in patients with vaginal cancer dispositioned to undergo surgery and bilateral lymph node dissection.

DETAILED DESCRIPTION:
The treatment of vaginal cancer is usually surgical removal of the vaginal tumor with removal of lymph nodes in the groin and/or pelvis. Patients who are not eligible to receive surgery usually receive radiation therapy.

Lymph nodes are a common site for the spread of vaginal cancer. Lymphatic mapping has been used in patients with other types of cancer to identify the "sentinel" lymph node. The sentinel lymph node is the lymph node believed to be at greatest risk for spread of the cancer. If the sentinel node does not contain cancer cells, then the remaining lymph nodes are almost always cancer free.

This research study will find out if the sentinel node concept can be applied to patients with vaginal cancer. The sentinel lymph node will be identified using a scan called "lymphoscintigraphy". A very small amount (less than one tenth of a teaspoon) of a radioactive material is injected around the edge of the tumor in the vagina, followed immediately by the scan. The scan is done in the Nuclear Medicine Department of M. D. Anderson before the patient has surgery or begins radiation therapy.

The dose of radiation injected into the vagina is much less than the dose received from a chest x-ray and therefore there are no special precautions needed after the injection. If the treatment plan is surgery, a second injection of the radioactive material may be necessary on the day of the operation because the radiation fades quickly. Patients who receive radiation therapy will not need a second injection. The radiation oncologist might use the information collected from the scan to help with treatment planning.

For patients having surgery, a special hand held instrument that measures radioactivity (similar to a Geiger counter) is used to help identify the location of the sentinel lymph node before and after the operation begins. Blue dye is also used to find the sentinel node. This requires the injection of up to a teaspoon of material called Isosulfan Blue around the tumor in the vagina. This is done while the patient is under anesthesia. The surgeon can then identify the sentinel node by its color (blue) and by its level of radioactivity (using the gamma counter).

Patients will be notified of the results of the mapping and lymphoscintigraphy during their hospitalization or their first clinic visit, depending on whether or not they had surgery.

This is an investigational study. Eighteen patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have invasive vaginal cancer, any histology, any stage.
* Patients with prior excision of the primary are eligible.
* Patients with recurrent vaginal cancer who have not had a prior inguinal or groin lymph node dissection.
* Patients undergoing either surgical resection and assessment of inguinal or groin lymph nodes, radiation therapy and/or chemotherapy.
* Patients must sign an IRB approved informed consent.

Exclusion Criteria:

* Known allergy to triphenylmethane compounds.
* Pregnancy.
* Prior radiation therapy to the vagina, vulva, groin or pelvis.
* Prior inguinal, femoral or pelvic lymphadenectomy.
* Patients who are not good surgical candidates.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2002-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Identification of sentinel lymph node(s) in patients with vaginal cancer using lymphoscintigraphy and intraoperative lymphatic mapping. | Preoperative and intraoperative, prior to radiation therapy, data collection

CONTACTS AND LOCATIONS:
Overall Officials: Charles Levenback, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Frumovitz M, Gayed IW, Jhingran A, Euscher ED, Coleman RL, Ramirez PT, Levenback CF. Lymphatic mapping and sentinel lymph node detection in women with vaginal cancer. Gynecol Oncol. 2008 Mar;108(3):478-81. doi: 10.1016/j.ygyno.2007.12.001. Epub 2008 Jan 10. PMID 18190952
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org